CLINICAL TRIAL: NCT00564473
Title: Use of Herbal Medicine Among Patients Hospitalized in a Department of Internal Medicine: A Cross-Sectional Survey
Brief Title: Use of Herbal Medicine in Internal Medicine Wards
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Dr. Noah Samuels, Shaare Zedek Medical Center
Other Study IDs: HERB.INTMED.08
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-10

CONDITIONS: Herb-drug Interactions
Keywords: internal medicine; herbal medicine; prevalence; attitudes; herb-drug interaction
MeSH Terms: conditions — Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: patients hospitalized in the Department of Internal Medicine of the Shaare Zedek Medical Center, Jerusalem, Israel.
  Interventions: Behavioral: questionnaire

INTERVENTIONS:
Behavioral: questionnaire — * questionnaire of demographic and medical data, use of and attituded toward herbal medicine.
  * Beck Depression Inventory-Second Edition (BDI-II)- Hebrew Translation

SUMMARY:
Herbs are physiologically active substances which can significantly affect the outcome of medical treatment, either by inhibiting or promoting drug disposition or through additive and synergistic effects when used in conjunction with conventional medications. Herb-drug interactions are potentially dangerous, and may be difficult to predict since regulation of the preparations is often lacking, and patients most often do not report the use of these products to their physicians. The risk for toxic effects and adverse interactions increases among high-risk groups, such as the elderly or patients with renal or hepatic disease. The purpose of this study is to study the prevalence of use of herbal medicine among patients hospitalized in the internal medicine department of an Israeli hospital, as well as examine the effect of herbal remedies on patient health, either beneficial or harmful. For this purpose, a questionnaire evaluating demographic data, medical history (both current and past), use of and attitudes towards herbal medicine will be administered to patients in the Department of Internal Medicine at the Shaare Zedek Medical Center in Israel. The Beck Depression Questionnaire will be used as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender
* Age 18 years and older

Exclusion Criteria:

* Neurological deficit or other medical condition precluding responding to the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized in a department of internal medicine
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
* prevalence of use of herbal medicine among patients hospitalized in the Department of Internal Medicine at the Shaare Zedek Medical Center in Jerusalem, Israel. | one year

SECONDARY OUTCOMES:
*prevalence of herb-drug interactions affecting treatment *rates of reporting use of herbal remedies *prevalence of toxic effects of herbal remedies *attitudes toward herbal medicine | one year

CONTACTS AND LOCATIONS:
Overall Officials: Noah Samuels, MD, Principal Investigator — Shaare Zedek Medical Center; Shoshanna Zevin, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel